CLINICAL TRIAL: NCT03727841
Title: Phase II Clinical Trial of Marizomib for Recurrent Low-Grade and Anaplastic Supratentorial, Infratentorial and Spinal Cord Ependymoma
Brief Title: Marizomib for Recurrent Low-Grade and Anaplastic Supratentorial, Infratentorial, and Spinal Cord Ependymoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The pharmaceutical company decided to close their program evaluating the study agent, Marizomib.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190011; 19-C-0011
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Anaplastic Ependymoma; Ependymoma; Ependymomas
Keywords: Proteasome Inhibitor; Penetration Across the Blood-Brain-Barrier (BBB); Apoptosis Induction; Targeted Therapeutic Effect; Tumor Progression
MeSH Terms: conditions — Ependymoma; Disease Progression | interventions — marizomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Arm 1 Marizomib (Experimental): Marizomib at days 1, 8, and 15 of each 28-day cycle
  Interventions: Drug: Marizomib
- P/Pregnancy Evaluation (No Intervention): Data collection on pregnancy, birth and Health of Child

INTERVENTIONS:
Drug: Marizomib — 0.8mg/m(2) intravenous (IV) on days 1, 8, and 15 of each 28-day cycle, 24 cycles total.
  Other Names: MRZ
  Arms: 1/Arm 1 Marizomib

SUMMARY:
Background:

Ependymomas are rare tumors that arise from the ependyma. That is a tissue of the central nervous system. They can develop in the brain or the spine. They are usually treated with surgery, radiation, and/or chemotherapy. Researchers want to see if the new drug marizomib can help people with a certain kind of ependymoma.

Objective:

To see if marizomib stops tumor growth and prolongs the time that the tumor is controlled.

Eligibility:

Adults age 18 and older who have been diagnosed with ependymomas and have already been treated with standard therapies

Design:

Participants will be screened with the following tests or recent results from similar tests:

* Medical history
* Physical exam
* Neurological assessment
* Electrocardiogram (EKG) to evaluate the heart
* Review of symptoms and ability to perform normal activities
* Computed tomographic scan (CT) or magnetic resonance imaging (MRI) to produce an image of the brain or spine.
* Blood and urine tests
* Tests of tumor samples. Participants may have to have new tumor samples taken.

Participants will get the study drug in cycles. Each cycle is 4 weeks. Participants will have up to 24 cycles.

Participants will get the study drug through a small plastic tube in a vein on days 1, 8, and 15 of each cycle.

During each cycle, some screening tests will be repeated.

Participants will answer questions about their general well-being and functioning.

About 4 5 weeks after finishing the study drug, participants will have a follow-up visit. They will answer questions about their health, get a physical and a neurological exam, and have blood tests. They may have an MRI or CT scan.

...

DETAILED DESCRIPTION:
Background:

* Ependymomas are rare primary brain tumors arising from radial glial stem cells. They comprise 5.2% of all pediatric primary brain tumors and 1.9% of all adult primary brain tumors.
* The standard therapy for newly diagnosed ependymoma is gross total resection followed by radiation therapy. For anaplastic ependymoma, recurrence rate is high with a median progression free survival (PFS) of 2.3 years.
* There are limited chemotherapy options for recurrent ependymomas, which have already been irradiated. Therefore, there is an unmet need to target novel pathways for treatment of ependymomas.
* About 70% of supratentorial ependymomas have a characteristic signature C11 orf95-V-Rel Avian Reticuloendotheliosis Viral Oncogene Homolog A (RELA) fusion which drives tumorigenesis in ependymomas by activating the nuclear factor kappa-light-chain-enhancer of activated B cells (NF-KB) transcription pathway.
* Marizomib is a second-generation irreversible proteasome inhibitor which penetrates across the blood-brain-barrier (BBB). It inhibits the activity of 20S proteasome in glioma cells, activates caspases, builds up reactive oxygen species and thus induces apoptosis. Marizomib blocks the NF-pathway by proteasome inhibition. Thus, it may have an additional targeted therapeutic effect in the RELA-fusion molecular subgroup of ependymomas.

Objective:

-To evaluate the efficacy of treatment with marizomib in RELA-fusion recurrent ependymoma and non RELA-fusion recurrent ependymoma as measured by progression-free survival at 6 months (PFS6).

Eligibility:

* Histologically proven intra-cranial or spinal ependymoma.
* Radiographic evidence of tumor progression
* Patients must be greater than or equal to 18 years old.

Patients must have had prior radiotherapy.

Design:

* This is a phase II study to determine the efficacy of marizomib in recurrent ependymoma.
* A novel 2-stage sequential design will be employed to conduct the trial for recurrent ependymoma.
* In the first stage, we will enroll 18 patients with RELA-fusion ependymoma and if 4 or more patients in Cohort 1 are progression free at 6 months, we will proceed to stage 2; otherwise, we will terminate the trial and conclude that marizomib is not effective.
* In the second stage, we will enroll 32 patients with non RELA-fusion ependymoma.
* Patients will be treated with marizomib in cycles consistent of 28 days until disease progression or a maximum of 24 cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Stage 1 Eligibility (Cohort 1 and 2)

Cohort 1

* Histologically confirmed by National Cancer Institute (NCI) Laboratory of Pathology intra-cranial or spinal V-Rel Avian Reticuloendotheliosis Viral Oncogene Homolog A (RELA)- fusion ependymoma of grade I, II or III.
* Has received two or fewer prior chemotherapy regimens

Cohort 2

* Histologically confirmed by NCI Laboratory of Pathology intra-cranial or spinal RELA-fusion ependymoma of grade I, II or III.
* Has received more than two prior chemotherapy regimens

  * Stage 2 Eligibility (Cohorts 3 and 4)

Cohort 3

* Histologically confirmed by NCI Laboratory of Pathology intra-cranial or spinal non RELA-fusion ependymoma of grade I, II or III.
* Has received two or fewer prior chemotherapy regimens

Cohort 4

* Histologically confirmed by NCI Laboratory of Pathology intra-cranial or spinal non RELA-fusion ependymoma of grade I, II or III.
* Has received more than two prior chemotherapy regimens.

  * Patients must have an evidence of tumor progression.
  * Patients must have had prior radiation therapy.
  * Patients must be greater than or equal to 18 years old. Currently, no dosing or adverse event data is available on the use of marizomib in patients < 18 years of age; therefore, only adults are included in this study. Patients < 18 years of age will be eligible for future pediatric trials.
  * Patients must have a Karnofsky performance status of greater than or equal to 60.
  * Patients must have adequate organ and marrow function as defined below:
  * leukocytes: greater than or equal to 3,000/microliters
  * absolute neutrophil count: greater than or equal to 1,500/microliters
  * platelets: greater than or equal to 100,000/microliters
  * hemoglobin: greater than or equal to 10 gm/dL (can be achieved by transfusion)
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT): less than or equal to 2.5 X institutional upper limit of normal
  * Bilirubin: <1.5 mg/dL
  * Creatinine up to 1.5-times upper institutional limits OR estimated glomerular filtration rate (eGFR) within normal as predicted by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (greater than or equal to 60 mL/min/1.73m(2).
  * Negative urine protein or urine protein concentration less than or equal to 60 mg/dL
  * The effects of marizomib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and up to 30 days after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Anticancer treatment within designated period of time before enrollment including:

  * surgery within 14 days
  * needle or core biopsy within 7 days
  * prior cytotoxic therapy within 28 days,
  * vincristine within 14 days
  * nitrosoureas within 42 days,
  * procarbazine administration within 21 days
  * non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid (radiosensitizer does not count) within 7 days; Avastin within 21 days. Any questions related to the definition of non-cytotoxic agents should be directed to the NCI Principal Investigator.
* Treatment with any investigational agent within 28 days before enrollment.
* History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless patient is in complete remission and off all therapy for that disease for a minimum of 3 years.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to marizomib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inadequately controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg).
* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
* New York Heart Association (NYHA) Grade II heart failure or greater or history of hospitalization for congestive heart failure diagnosis within 12 months prior to enrollment.
* History of myocardial infarction or unstable angina within 3 months prior to enrollment.
* A marked baseline prolongation of QT interval (QT)/corrected QT interval (QTc) (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Frederica's QT correction

formula.

* A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Current use of concomitant medications that prolong the QT/QTc interval
* History of stroke or transient ischemic attack within 3 months prior to enrollment.
* Pregnant women are excluded from this study because marizomibs potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with marizomib, breastfeeding should be discontinued if the mother is treated with marizomib.
* Patients receiving combination antiretroviral therapy for treatment of Human Immunodeficiency Virus (HIV) or active anti-viral treatment for Hepatitis A, B or C infection. Anti-viral therapy, when combined with marizomib, poses a potential for pharmacokinetic interactions. Marizomib also increases immunosuppression, placing patients at an increased risk of acquiring lethal infections. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Inclusion Criteria for Pregnancy Cohort (P)

Because the drug manufacturer would like to study the effect of the study therapy on pregnancy, and because the required information cannot be collected unless a subject is enrolled per ruling of the OGC, the following additional groups of subjects may be enrolled if necessary.

-A child whose parent (male or female) is/was an active participant in the study at any time during the childs gestation. Active participant is defined as having received at least one dose of study therapy through 6 months after the last dose of study therapy.

OR

* An expectant mother of child whose father is/was an active participant in the study at any time during the childs gestation. The father must have received at least one dose of study therapy. Active participant is defined as having received at least one dose of study therapy through 6 months after the last dose of study therapy.
* The expectant mother must be age 18 or older and must have the capacity to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Gilbert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
1. Biomedical Translational Research Information System (BTRIS): All IPD recorded in the medical record will be shared with intramural investigators upon request.
  2. Database of Genotypes and Phenotypes (dbGaP): All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: BTRIS: Clinical data available during the study and indefinitely. dbGaP: Genomic data are available once genomic data are uploaded per protocol genomic data sharing (GDS) plan for as long as database is active.
Access Criteria: BTRIS: Clinical data will be made available via subscription to BTRIS and with the permission of the study principal investigator (PI).
  dbGaP: Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Wu J, Armstrong TS, Gilbert MR. Biology and management of ependymomas. Neuro Oncol. 2016 Jul;18(7):902-13. doi: 10.1093/neuonc/now016. Epub 2016 Mar 28. PMID 27022130
- [Background] Harrison SJ, Mainwaring P, Price T, Millward MJ, Padrik P, Underhill CR, Cannell PK, Reich SD, Trikha M, Spencer A. Phase I Clinical Trial of Marizomib (NPI-0052) in Patients with Advanced Malignancies Including Multiple Myeloma: Study NPI-0052-102 Final Results. Clin Cancer Res. 2016 Sep 15;22(18):4559-66. doi: 10.1158/1078-0432.CCR-15-2616. Epub 2016 Apr 26. PMID 27117181
- [Background] Di K, Lloyd GK, Abraham V, MacLaren A, Burrows FJ, Desjardins A, Trikha M, Bota DA. Marizomib activity as a single agent in malignant gliomas: ability to cross the blood-brain barrier. Neuro Oncol. 2016 Jun;18(6):840-8. doi: 10.1093/neuonc/nov299. Epub 2015 Dec 17. PMID 26681765
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0011.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were plans to enroll participants in the pregnancy arm, however, participants were unable to be reached, thus no participants were enrolled on this arm, and no data was collected.
Groups:
- 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies: Marizomib at days 1, 8, and 15 of each 28-day cycle
  Marizomib: 0.8mg/m(2) intravenous (IV) on days 1, 8, and 15 of each 28-day cycle, 24 cycles total.
  Participants with Intra-cranial or Spinal V-Rel Avian Reticuloendotheliosis Viral Oncogene Homolog A (RELA)-fusion Ependymoma who have had none, 1 or 2 prior chemotherapies.
- 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies: Participants with intra-cranial or spinal RELA-fusion ependymoma who had more than two prior chemotherapies.
Period: Overall Study
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (13.8) | 32.3 (0) | 43.63 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Are Progression-free at 6 Months Time Point After Initiation of Treatment
Description: Progression was assessed by the Response assessment in neuro-oncology criteria (RANO) and is defined as a 25% increase in the sum of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline. Appearance of new lesions, or clear worsening of any evaluable disease. Failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0

2. Secondary Outcome: Number of Toxicities by Grade Using the Common CTCAE Version 5.0.
Description: To determine the safety of marizomib in recurrent ependymoma patients and in a subset of patients with more than 2 prior chemotherapies (RELA-fusion Cohort 2 and non-RELA-fusion Cohort 4).
Time Frame: At end of study, up to 16 months
Measure: Number; unit: Toxicities
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Toxicities
  Grade 1 | 35 | 13
  Grade 2 | 24 | 5
  Grade 3 | 6 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

3. Secondary Outcome: Number of Participants That Have Progressive Disease After 6 Months
Description: To estimate the efficacy of marizomib in recurrent ependymoma patients (RELA- fusion Cohort 2 and non RELA-fusion Cohort 4) with more than 2 prior chemotherapies as measured by progression free disease after 6 months. Progression was assessed by the Response Assessment in Neuro-oncology (RANO) criteria and is defined as a 25% increase in the sum of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline. Appearance of new lesions, or clear worsening of any evaluable disease. Failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Population: The one participant in Cohort 2 had progressive disease prior to 6 month mark and we did not enroll in Cohort 4 due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With 12-month Progression-free Survival (PFS12)
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

5. Secondary Outcome: Symptom Severity Using the MD Anderson Symptom Inventory- Brain Tumor (MDASI-BT) and/or MD Anderson Symptom Inventory - Spine Tumor Module (MDASI-SP) Instrument
Description: Changes in quality of life using the MD Anderson Symptom Inventory- Brain Tumor (MDASI-BT) and/or MD Anderson Symptom Inventory - Spine Tumor Module (MDASI-SP) instrument was used to determine symptom severity.To longitudinally evaluate participant reported outcome measures using self-reported symptom severity with daily activities using the MDASI-BT and/or MDASI-SP instrument.
Time Frame: End of study
Population: This outcome measure was not done because we were unable to determine due to low accrual and few data timepoints for which meaningful data could be extracted.
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Assessed Using the Response Assessment in Neuro-oncology Criteria (RANO) for Complete Response (CR) + Partial Response (PR)
Description: To estimate the efficacy of marizomib in recurrent ependymoma patients (RELA- fusion Cohort 2 and non RELA-fusion Cohort 4) with more than 2 prior chemotherapies as measured by objective response. Complete Response is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Partial Response is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
Time Frame: Up to 16 months
Population: We did not enroll to Cohort 4 due to early termination of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

7. Secondary Outcome: Median Amount of Time Subject Survives 12 Months After Therapy
Description: Median amount of time subject survives 12 months after therapy
Time Frame: 12 months after therapy
Population: This outcome measure was not done. We were unable to determine as participants were taken off study for early study termination prior to the 12 months post therapy timepoint.
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival (OS) of RELAfusion and Non RELA-fusion Recurrent Ependymoma Patients Treated With Marizomib.
Description: OS is defined as the time from treatment start date until date of death or date last known alive.
Time Frame: Start of treatment until end of study
Population: This outcome measure was not done. We were unable to determine for non RELA-fusion recurrent ependymoma patients since we did not enroll in those cohorts due to early study termination. And for the 4 participants with RELA-fusion recurrent ependymoma enrolled, the study was prematurely terminated pharmaceutical sponsor.
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Symptom Interference Using the MD Anderson Symptom Inventory- Brain Tumor (MDASI-BT) and/or MD Anderson Symptom Inventory - Spine Tumor Module (MDASI-SP) Instrument
Description: Changes in quality of life using the MD Anderson Symptom Inventory- Brain Tumor (MDASI-BT) and/or MD Anderson Symptom Inventory - Spine Tumor Module (MDASI-SP) instrument was used to determine symptom interference.To longitudinally evaluate participant reported outcome measures using self-reported symptom interference with daily activities using the MDASI-BT and/or MDASI-SP instrument.
Time Frame: End of study
Population: as for outcome 5
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 27 days, and 7 months and 22 days for the first and second group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
Number analyzed (Participants) | 3 | 1
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 14 months and 27 days, and 7 months and 22 days for the first and second group respectively.
Arm/Group | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies (N=3) | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies (N=1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Cohort 1 - Participants With Ependymoma Who Had None, One or Two Prior Chemotherapies (N=3) | 2/Cohort 2 - Participants With Ependymoma Who Had More Than Two Prior Chemotherapies (N=1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (7) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 1 (3)
Nausea (Gastrointestinal disorders) | 3 (9) | 1 (3)
Nervous system disorders - Other, Aphasia (word-finding difficulties) (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (5) | 1 (5)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (6) | 0 (0)
White blood cell decreased (Investigations) | 1 (5) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03727841/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03727841/ICF_001.pdf